CLINICAL TRIAL: NCT02891213
Title: Study of the Role of Soluble Forms of RAGE (sRAGE/esRAGE) as Diagnostic and Prognostic Biomarkers of Systemic Lupus Erythematosus.
Acronym: R-PA14098
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA14098
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Lupus Erythematosus

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- LE (Lupus Erythematosus) group: * Samples of the LE (Lupus Erythematosus) group from a specimen collection : "Lupus BioBanque du Rhin Supérieur" (LBBR UF 9882).
  * It's a historical cohort of lupic patients which samples have been collected from many centers in France and Germany and stored in a biobank "Lupus BioBanque du Rhin Supérieur" (project : LBBR UF 9882).

SUMMARY:
Systemic Lupus Erythematosus (SLE) is the most common systemic autoimmune disease. The clinical manifestations are severe and affect multiple target organs such as the kidney, central nervous system, skin, heart and joints. Despite the progress made in the therapeutic approach with new immunosuppressive regimens, morbi-mortality is still high. Therefore, it's important to identify new biomarkers to help clinicians to predict severity and evolution of the disease for better adaptation of treatments and try to improve the prognosis.

RAGE (Receptor for Advanced Glycation Endproducts) :

RAGE (Receptor for Advanced Glycation Endproducts) is an ubiquitous membrane receptor, involved in development of many diseases such as diabetes, chronic renal failure but also in vascular remodelling, inflammatory, infectious deseases and cancer. RAGE regulates a number of crucial cell processes like inflammation, and tissue and cellular homeostasis.

RAGE is able to bind not only the advanced glycation end products (AGEs) such as pentosidine, carboxymethyllysine (CML), methyl-glyoxal-hydroimidazolone-1 (MG- H1), but also other ligands such as HMGB1 (high mobility group box1), and S100A8/A9 proteins which have been correlated in recent studies to the activity index of SLE. The activation of RAGE leads to a cascade of intracellular signaling and activation of the transcription factor NF-ΚB . NF-ΚB enable the traduction of proinflammatory cytokines such as IL-6, IL-1α ,IFN-γ. In SLE, these cytokines involved in perpetuation of inflammation and tissue damages including lupus nephritis. Moreover, the activation of RAGE induces the expression of adhesion molecule such as sICAM -1 and sVCAM -1 wich were recently involved in SLE vasculitis.

Soluble forms of RAGE, sRAGE and esRAGE :

RAGE is a proinflammatory membrane receptor. But RAGE also exists in soluble plasma forms, esRAGE (secreted form) and sRAGE (a truncated form as cleaved by MMP9 and ADAM10 enzymes). esRAGE and sRAGE have the same ligand-binding specificity as RAGE and may function as a 'decoy receptor' by binding pro-inflammatory ligands and preventing them from accessing cell surface RAGE (Kierdorf and Fritz, 2013). Therefore, both soluble forms have an anti-inflammatory action. Several studies have shown a decrease in circulating levels of sRAGE in patients with Rheumatoid Arthritis, or Sjögren Syndrome compared with healthy controls. However, the role of RAGE in SLE remains unknown.

RAGE and Systemic Lupus Erythematosus, recent advances :

Our team (Laboratory of Nephrology, CNRS UMR 7369, URCA) showed in a study in lupus RAGE knockout mice (B6/ MRL-FAS lpr/J RAGE-/-) a strong involvement of RAGE in systemic manifestations SLE. Recently, another report showed that sRAGE has an anti-inflammatory effect on the lupus nephritis and could be a potent therapy in mice.

In humans, two studies show a correlation between the plasma level of sRAGE and lupus phenotype ( Nienhuis et al. , 2008).

Working hypothesis :

Based on the results and those of the current studies, the investigators think that RAGE axis and its soluble forms play a crucial role in the complex pathogenesis of SLE.

The investigators hypothesize that plasma levels sRAGE and esRAGE are a reflection of the activity and the development of SLE in humans. Soluble forms of RAGE and ligands may be novel biomarkers of SLE and sRAGE a potent therapeutic target.

DETAILED DESCRIPTION:
Expected results :

The investigators expect a correlation between serum sRAGE, esRAGE and activity of SLE and the presence of visceral involvement. Furthermore this study will allow us to analyze for the first time in a lupus population, the correlation between soluble forms of RAGE (esRAGE, sRAGE) and cytokines and molecules involved in lupus visceral involvement as IL-6, IL-1α, IFN-γ, sICAM-1 and sVCAM-1.

Completion of our project, will allow better understanding of the role of RAGE and RAGE ligand in SLE activity and will provide rationale for prospective study.

Future perspectives will include assessment of the risk-benefit for the use of anti-RAGE strategies or recombinant sRAGE/esRAGE molecules as adjuvant treatment for SLE.

Study Design : the investigators designed an retrospective, analytic, transversal, mulitcentric study. the investigators would like to use the serum and the clinical information collected in "Lupus BioBanque du Rhin Supérieur" (LBBR UF 9882) to measure soluble forms of RAGE, RAGE-ligands, cytokines, and sICAM and sVCAM. The investigators would like to include 150 patients in this study.

Aim 1: The main objective of this study is to investigate the association between Systemic Lupus Erythematosus (SLE) activity as measured by the SLEDAI score and serum concentrations of sRAGE and esRAGE.

Aim 2 : The study of the correlation between the activity of other activity markers of SLE and soluble forms of RAGE :

1. the concentration of RAGE ligands (AGEs like CML, pentosidine and MG-H1) and soluble forms of RAGE (esRAGE, sRAGE)
2. the cytokine profile (IL-6, IL-1α, IFN-γ) and soluble forms of RAGE (esRAGE, sRAGE)
3. The concentrations of sICAM-1 and sVCAM-1 and soluble forms of RAGE (esRAGE, sRAGE)

Methods :

Inclusion criteria are :

* the LBBR inclusion criteria
* and Absence of immunomodulatory treatment,
* and preserved renal function (MDRD> 60ml/min).

Exclusion criteria are :

* renal failure defined by MDRD clearance < 60 mL/min/m2,
* or neoplasia,
* or diabetes,
* or other autoimmune disease,
* or current immunosuppressive treatments.

Data collection : About 500 μl of serum will be necessary for each patients to make all measurements.

Mass spectrometry will be used for measurement of RAGE ligands (Advanced glycation end products such as CML, pentosidine and MG-H1).

Commercially available ELISA kits will be used for measurement of sRAGE, esRAGE, sVCAM1.

Flow Cytometry will be used for measurement of cytokines (IL-6, IL-1a, IFN-y) and sICAM1.

ELIGIBILITY:
Inclusion Criteria:

* patients have been included in the LBBR biobank
* absence of immunomodulatory treatment,
* preserved renal function (MDRD> 60ml/min).

Exclusion Criteria:

* renal failure defined by MDRD clearance < 60 mL/min/m2,
* neoplasia,
* diabetes,
* other autoimmune disease,
* current immunosuppressive treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is the cohort of lupic patients have been included in "Lupus BioBanque du Rhin Supérieur".
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
concentration of RAGE ligands | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France